CLINICAL TRIAL: NCT01413984
Title: Substance Abuse and Trauma in Incarcerated Women: An Effectiveness Study
Brief Title: Substance Abuse and Trauma in Incarcerated Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tulsa (Other)
Responsible Party: Principal Investigator, Rachael Swopes, Graduate Student, University of Tulsa
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TU 11-18
Record Dates: First submitted 2011-08-03; First posted 2011-08-10 (Estimated); Last update posted 2014-03-18 (Estimated); Status verified 2014-03

CONDITIONS: Substance Abuse; Trauma; Post Traumatic Stress Disorder; Integrated Treatment; Incarcerated Women
Keywords: Trauma; incarceration; treatment; substance abuse
MeSH Terms: conditions — Substance-Related Disorders; Wounds and Injuries; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cognitive behavioral group treatment (Experimental): Helping Women Recover/Beyond Trauma integrated substance abuse and trauma treatment group. (Dr. Covington)
  Interventions: Behavioral: Helping Women Recover/Beyond Trauma
- comparison group (No Intervention): a comparison group of incarcerated women will receive the pre and post assessments with no interventions.

INTERVENTIONS:
Behavioral: Helping Women Recover/Beyond Trauma — Four treatment rounds will be conducted, and a goal of 20 women (10 from each group) will be recruited to participate in each round. A new treatment group will start every four months. Sessions are approximately 2 hours each, 3-4 times per week over four months in a group format. This treatment program will focus on the integrated treatment of trauma and substance abuse in women. Versions of the curriculum exist both for community and corrections populations. In this intervention the corrections version will be used.
  Arms: cognitive behavioral group treatment

SUMMARY:
The proposed study will evaluate Covington's Helping Women Recover (HWR) plus Beyond Trauma (BT) curriculum with female offenders at Eddie Warrior Correctional Facility in Taft, Oklahoma. The purpose of the proposed study is to expand previous findings by including a comparison group of women that are not receiving treatment but are otherwise eligible, and by using outside evaluators to conduct the assessments. Furthermore, this study will extend the outcomes measured in previous evaluations by including measures of sleep disturbance, posttraumatic cognitions, and a more extensive assessment of trauma-related symptoms. The hypotheses for this study are listed below:

1. Incarcerated women with substance use disorders and history of trauma enrolled in the integrated treatment program (HWR plus BT) will report significantly fewer symptoms on measures of posttraumatic stress and associated cognitions, substance use, depression, and related symptoms following treatment than those in the comparison group.
2. Those in the treatment group will improve significantly more than those in the comparison group on the symptoms listed above.

ELIGIBILITY:
Inclusion Criteria:

* Incarcerated women at Eddie Warrior Correctional Center (EWCC) in Taft, Oklahoma
* The following 6 criteria are then employed at EWCC for HWR/BT treatment eligibility:

  1. An Level of Service Inventory (LSI) score of 30 or greater
  2. An LSI protective score of 15 or less
  3. 1.5 years or less remaining in prison
  4. A Case Plan identifying substance abuse treatment need
  5. Ability to read and comprehend
  6. 18 years of age or older

Exclusion Criteria:

* Under age 18
* Not incarcerated
* More than 1.5 years remaining in prison
* LSI score less than 30 or a protective of more than 15
* No identified substance abuse need
* Inability to read and comprehend

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2010-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
PTSD checklist (change from baseline at one week post treatment) | one-week before treatment, one week post treatment
  17 item post traumatic stress disorder symptoms checklist will be administered pre treatment and one week following 4 month treatment completion.
Trauma Related Nightmare Survey (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  brief assessment of nightmare frequency and severity to be administered pre-treatment and one week following 4 month treatment completion.
Posttraumatic Cognitions Inventory (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  36 item assesment of cognitions related to world, self and blame to be administered pre-treatment and one week following 4 month treatment completion.
CES-D, NIMH (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  Center for Epidemiologic Studies Depression Scale (CES-D), NIMH is a 20 item depression inventory to be administered pre-treatment and one week following 4 month treatment completion.
Drug-Taking Confidence Questionnaire (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  50 item assessment of alcohol and drugs self efficacy to be administered pre-treatment and one week following 4 month treatment completion.
Trauma Symptoms Inventory (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  100 item trauma symptoms questionnaire to be administered pre-treatment and one week following 4 month treatment completion.

SECONDARY OUTCOMES:
Parenting Stress Index for Incarcerated Women (change from baseline at one week post treatment) | one week before treatment, one week post treatment
  two scales from the PSI and selected parenting issues from incarcerated women to be administered pre-treatment and one week following 4 month treatment completion.

CONTACTS AND LOCATIONS:
Overall Officials: Rachael Swopes, M.S., Principal Investigator — University of Tulsa
Locations (1):
- Eddie Warrior Correctional Facility, Taft, Oklahoma, United States